CLINICAL TRIAL: NCT06717750
Title: A Single-arm, Open-label, Single/Multiple-dose Escalation, and Cohort Expansion Phase Ia/Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of Oral CSCJC3456 Tablets in Patients With Advanced Malignant Solid Tumors
Brief Title: A Study of CSCJC3456 in Patients With Advanced Malignant Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Changshan ConjuChem BioPharmaceutical Research and Development (Hebei) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSCJC CA101
Record Dates: First submitted 2024-11-26; First posted 2024-12-05 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Advanced Malignant Solid Tumors
Keywords: Neoplasms; Antineoplastic Agents; Tyrosine Kinase Inhibitors; Protein Kinase Inhibitors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CSCJC3456 monotherapy (Experimental): * Phase Ia: Single and Multiple Dose Escalation.
  * Phase Ib: Cohort Expansion.
  Interventions: Drug: CSCJC3456 tablet

INTERVENTIONS:
Drug: CSCJC3456 tablet — * Phase Ia: Single and Multiple Dose Escalation.
    1. Dosage form: tablet.
    2. Dosage: 7 dose groups, 5 mg, 15 mg, 30 mg, 45 mg, 60 mg, 80 mg, 100 mg.
    3. Frequency: once daily (tentative), or twice daily and other options (adjusted based on the results of the preliminary trials).
    4. Duration: 5 mg(days 1-28; 28 days per cycle), other groups (days 1-14; 21 days per cycle) .
  * Phase Ib: Cohort Expansion. Dosage and dosing regimen: according to the recommended dosage and dosing cycle from the Phase Ia study.

SUMMARY:
This study is a multicenter, open phase I clinical study of dose escalation, cohort expansion study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of CSCJC3456 in patients with advanced malignant solid tumors.

DETAILED DESCRIPTION:
CSCJC3456 is a multi-target tyrosine kinase inhibitor, and this is the first-in-human trial of CSCJC3456. This study adopts an open-label, non-randomized, single-arm, dose-escalation, and cohort expansion research design, and is divided into two parts, Phase Ia and Phase Ib.

Phase Ia is a single and multiple dose escalation trial with an open-label design, aiming to evaluate the safety, tolerability, PK, and PD characteristics of CSCJC3456 tablets, preliminarily assess the anti-tumor efficacy, and recommend the dose for Phase Ib study.

Phase Ib is a single-arm cohort expansion study conducted in participants with four target solid tumors, based on the recommended dosage and dosing cycle from the Phase Ia study. The actual tumor types for the Phase Ib study will be adjusted according to the safety and efficacy data from the Phase Ia study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and follow protocol requirements;
2. Aged 18 to 75 (both inclusive), male or female, regardless of race;
3. Expected survival period ≥ 12 weeks;
4. ECOG PS score ≤1;
5. Phase Ia study:

   ● Participants with advanced malignant solid tumors confirmed by pathology or cytology, who have experienced disease progression despite standard treatment, are intolerant to standard treatment, or lack effective standard treatment; and who possess at least one measurable lesion in accordance with RECIST v1.1 criteria;

   Phase Ib study:
   * Cohort A (hepatocellular carcinoma, including at least 2 participants with FGFR4 positivity), Cohort B (colorectal cancer, including at least 2 participants with FGFR1 or FGFR2 positivity), Cohort C (gastric cancer (including adenocarcinoma at the gastroesophageal junction), including at least 2 participants with FGFR1 or FGFR2 positivity), Cohort D (recurrent/metastatic endometrial cancer, including at least 2 participants with FGFR2 or FGFR3 positivity), or other sensitive tumor types identified in phase Ia trial, confirmed by histology or cytology, who have failed or are intolerant to standard treatment. Investigators may adjust participant selection based on their response to treatment in the trial and communication with the sponsor.
   * Each cohort of participants had at least one measurable lesion that met the criteria of RECIST v1.1.
6. Before the first dose, the participant has recovered from the toxic effects of the previous last treatment (CTCAE grade ≤ 1, except for special conditions such as "hair loss" and "pigmentation"), and in addition, the investigator judges that the corresponding AE did not pose a safety risk;
7. Systolic blood pressure ≤150 mmHg, diastolic blood pressure ≤90 mmHg, and no changes in antihypertensive medication and dosage within 7 days prior to the first administration.
8. Adequate Organ and bone marrow function.
9. Female participants of childbearing age must undergo a serum pregnancy test 7 days before starting the study medication, and the result must be negative. They must also be willing to adopt a medically approved highly effective contraceptive measure (e.g., an intrauterine device, contraceptive pills, or condoms) during the study period and for 3 months after the last administration of study medication. Male participants whose partners are female of childbearing age should agree to adopt an effective contraceptive method during the study period and for 3 months after the last administration of study medication. Breastfeeding women should agree to cease breastfeeding during the study period and for 3 months after the last administration of study medication.
10. Have the gene sequencing results of the current tumor, or are willing to provide tumor tissue specimens (paraffin-embedded tissue blocks, or serial sections).

    * Specimens are preferably derived from recently collected and usable tumor tissues. For relevant instructions, please refer to the Central Laboratory Manual.
    * In cases where there is insufficient tumor tissue (e.g., insufficient number of available slides, including situations where no tissue specimens are available) and the investigator believes that another tumor tissue biopsy is unsafe, intolerable, infeasible, or the patient refuses, the patient can be enrolled in the study after discussion with the sponsor.

Exclusion Criteria:

1. Previous or current diagnosis of other types of malignancy, except for the following:

   1. Radically cured basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, cervical carcinoma in situ, or breast cancer in situ;
   2. Second primary cancer that has been cured with no recurrence within 5 years;
2. Patients who are allergic to any component of the study drug or have a history of severe allergies;
3. Having received any of the following treatments or medications before the first study treatment:

   1. Major surgery or major trauma occurred within 4 weeks before the first study drug, but diagnostic tissue biopsies are allowed. Severe trauma refers to unhealed wounds, ulcers, or fractures;
   2. Received treatment with traditional Chinese patent medicines and simple preparations with anti-tumor indications within 2 weeks before the first study drug treatment;
   3. Received anti-neoplastic therapies (including chemotherapy, radiotherapy, immunotherapy, targeted therapy, biologic therapy, or tumor embolization) within 4 weeks or 5 half-lives of the investigational drug prior to the first dose, whichever is shorter;
   4. Have received a potent CYP2C8 or CYP3A4 inducer within 2 weeks before the first dose; Or have received potent CYP2C8 or CYP3A4 inhibitors with less than 5 half-lives before the first dose;
   5. Have received medications known to significantly prolong the QT interval (e.g., class Ia and class III antiarrhythmic drugs) within 1 week or 5 half-lives of the investigational drug prior to the first dose, whichever is shorter;
   6. Previously received treatment with FGFR inhibitors (e.g., pemetrexed, erdafilone, infigranib, forodesine, ponatinib, dovitinib, nintedanib, AZD4547, NVP-BGJ398, LY2784455, BAY1163877, etc.);
4. Patients with a history of central nervous system metastasis or spinal cord compression. Those who meet the following criteria can be enrolled:

   1. Patients who have clearly received treatment and have been clinically stable for 4 weeks after discontinuing anticonvulsants and steroids prior to the first administration of the study drug (definition of clinical stability: no clinical accompanying symptoms such as intracranial hypertension or neurological symptoms within 4 weeks, and imaging findings indicating stable lesions within 4 weeks prior to the first administration of the drug);
   2. For patients with brain metastases, ≥21 days from whole brain radiation therapy (WBRT) to the first study treatment administration, ≥7 days from stereotactic radiosurgery (SRS) to the first study treatment administration, or ≥28 days from surgical resection to the first study treatment administration;
5. Advanced patients who have symptoms, spread to viscera, and are at risk of life-threatening complications in a short period of time, patients who have undergone at least two paracentesis and drainage within 4 weeks before the first dose, or patients who have undergone one paracentesis and drainage but have unstable pleural effusion, peritoneal effusion, or pericardial effusion;
6. Within the 6 months prior to screening, having a cardiovascular disease.
7. Uncontrolled systemic diseases, such as diabetes, hypertension, etc.;
8. Currently suffering from sudden pulmonary disease, interstitial lung disease or pneumonia, pulmonary fibrosis, acute pulmonary disease, etc., except for local interstitial pneumonia induced by radiotherapy;
9. Patients with a clear tendency towards gastrointestinal bleeding, including the following conditions: those with a history of black stool or hematemesis within 2 months; those whom investigators believe may have a high risk of major gastrointestinal bleeding;
10. Patients with previous or current grade ≥3 gastrointestinal perforation or visceral fistula;
11. Grade ≥3 diarrhea during the screening period;
12. Evidence of active infection.
13. Positive for human immunodeficiency virus (HIV RNA) or treponema pallidum antibodies;
14. Have multiple factors that affect oral medication (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.) or a condition that the investigator has judged to severely affect gastrointestinal absorption;
15. Having a clear history of neurological or psychiatric disorders, including epilepsy or dementia;
16. Having received any investigational drug within 4 weeks before the first administration, or participating in another clinical study at the same time (excluding the following situations: the patient is participating in an observational, non-interventional clinical study, or is in the follow-up period of an interventional clinical study; or the last study drug has been taken for more than 5 half-lives);
17. Patients deemed unsuitable for inclusion in this study by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ia: Dose Limiting Toxicity (DLT) | From first dosing at cycle 0 to the end of cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Number and proportion of individuals experiencing DLT. According to the NCI-CTCAE V5.0 toxicity evaluation criteria, DLT is defined as a certain level of toxicity related to the study drug (including definitely related, probably related, and possibly related) occurring during the first treatment cycle (C0D1~C1D21) of single and multiple administrations.
Phase Ia: Maximum Tolerated Dose (MTD) | From first dosing at cycle 0 to the end of cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  MTD is defined as the maximum dose at which the number of cases with DLT is ≤1/6 during the DLT observation period. To determine MTD, 6 evaluable participants are required.
Phase Ia: Assessment of safety and toxicity profile | From enrollment until the 28 days after the last study dose.
  Number of participants who experienced AEs, SAEs, and changes in physical examination, vital signs, ECOG score, imaging examination, laboratory tests, and 12-lead electrocardiogram, etc.
Phase Ib: Objective Response Rate (ORR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  ORR is defined as the proportion of participants whose tumors have achieved complete response (CR) and partial response (PR) after treatment, with response confirmed at least 4 weeks after the first assessment of CR or PR.

SECONDARY OUTCOMES:
Phase Ia and Phase Ib: Terminal Phase Half-life (t1/2 ) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia and Phase Ib: Maximum plasma concentration (Cmax) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia and Phase Ib: Time to reach Cmax (tmax) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia and Phase Ib: Area Under the Curve (AUC) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia and Phase Ib: Apparent Volume of Distribution (Vz/F) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia and Phase Ib: Apparent Clearance Rate (CL/F) | From enrollment to the end of cycle 1, phase Ia includes cycles 0 and 1, while phase Ib includes cycle 1. Cycle 0 has 3 days, and cycle 1 has 21 days.
  Evaluate drug concentration-time data by individual subject for single or repeated dosing of CSCJC3456.
Phase Ia: Objective response rate (ORR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  ORR is defined as the proportion of participants whose tumors achieve complete response (CR) or partial response (PR) after treatment.
Phase Ia and Phase Ib: Disease control rate (DCR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  DCR is defined as the proportion of participants whose tumors achieve complete response (CR), partial response (PR), or stable disease (SD) after treatment.
Phase Ia and Phase Ib: Durable objective response (DOR) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  DOR is defined as the period from the start of objective response recorded to the first occurrence of tumor progression or death due to any cause.
Phase Ia and Phase Ib: Progression-free survival (PFS) | From enrollment to the date of first documented progression or death due to any cause, whichever came first (up to approximately 2 years).
  PFS is defined as the time period from the initiation of treatment to the occurrence of tumor progression or death due to any cause.
Phase Ib: Overall survival (OS) | From enrollment to the date of death due to any cause (up to approximately 2 years).
  OS is defined as the time from the initiation of treatment to death due to any cause.
Phase Ib: Assessment of safety and toxicity profile | From enrollment until the 28 days after the last study dose.
  Number of participants who experienced AEs, SAEs, and changes in physical examination, vital signs, ECOG score, imaging examination, laboratory tests, and 12-lead electrocardiogram, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, M.D., Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The First Hospital of China Medical University, Shenyang, Liaoning

IPD SHARING:
Plan to Share IPD: No